CLINICAL TRIAL: NCT04121559
Title: A Feasibility Study of Delivering Adolescent Nutrition Interventions Through School-Based Platforms in Ethiopia: A Cluster-Randomized Evaluation
Brief Title: A Feasibility Study of Delivering Adolescent Nutrition Interventions Through School-Based Platforms in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Addis Continental Institute of Public Health (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHND-19-0949
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Dietary Diversity
Keywords: Adolescent Nutrition; Ethiopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A&T intervention areas: adolescent-nutrition-focused behavior change interventions delivered through government primary schools and communities
  Interventions: Behavioral: School Interventions; Behavioral: Community Interventions; Behavioral: School System Interventions
- Control (No Intervention): Comparison areas: standard activities at government primary schools

INTERVENTIONS:
Behavioral: School Interventions — 1. Classroom lessons on nutrition, dietary diversity, healthy food choices and handwashing.
  2. Principals provide messages on nutrition, dietary diversity, healthy food choices and handwashing at flag events or school assemblies.
  3. Selected adolescent girls are mentored by science teachers as peer mentors and hold weekly group discussions with other girls to discuss nutrition, dietary diversity, healthy food choices and handwashing.
  4. Trained science teachers take anthropometric measurements of adolescent girls to calculate BMI and provide nutrition counseling.
  5. Parent-teacher meetings to inform and encourage parents about adolescent nutrition, dietary diversity, healthy snacks, and handwashing.
  Arms: Intervention
Behavioral: Community Interventions — 1. Home visits by HEWs and/or community volunteers to discuss with parents about adolescent nutrition, dietary diversity, healthy food choices, and handwashing.
  2. Community gatherings by HEWs and meetings with religious leaders to discuss with parents about adolescent nutrition, dietary diversity, healthy food choices, and handwashing.
  Arms: Intervention
Behavioral: School System Interventions — 1. Workshop on the adolescent nutrition interventions for school principals, science teachers, HEWs, supervisors, and woreda officers.
  2. Biweekly supportive supervision on adolescent nutrition activities for schools and HEWs by school supervisors or woreda health/education office.
  Arms: Intervention

SUMMARY:
Alive & Thrive (A&T) is an initiative that supports the scaling up of nutrition interventions to save lives, prevent illnesses, and contribute to healthy growth and development through improved maternal nutrition, breastfeeding and complementary feeding practices. In Ethiopia, A&T tested the feasibility of implementing a package of locally tailored adolescent nutrition interventions through school-based (flag assemblies, classroom lessons, girls' clubs, peer mentoring, weight and height measurement, and parent-teacher meetings) and community platforms (health post and home visits and community gatherings). The evaluation used a two-arm cluster-randomized, non-masked trial design, consisting of two cross-sectional surveys in 2019 and 2021.

DETAILED DESCRIPTION:
Adolescence is a critical period of physical and psychological development and for achieving human potential. Rapid physical, psychosocial and cognitive growth and development is coupled with increased energy and nutrient requirements (Das et al., 2017; Spear 2002). Poor nutrition during adolescence can have adverse consequences impacting health in adulthood. The significance of nutrition during adolescence is especially important for girls, as poor nutrition can affect their well-being as well as the survival, health and well-being of their children (Das et al. 2017).

A&T Ethiopia implemented a package of adolescent nutrition interventions through school-based (flag assemblies, classroom lessons, girls' clubs, peer mentoring, weight and height measurement, and parent-teacher meetings) and community platforms (health post and home visits and community gatherings). IFPRI tested the feasibility of the behavior-change interventions and examined their impacts on adolescent girls' diets, compared with standard school and community activities in control areas.

The evaluation used a two-arm cluster-randomized, non-masked trial design, consisting of two cross-sectional surveys of in-school adolescent girls aged 10-14 years enrolled in grades 4-8. The unit of randomization is the primary school which includes grades 1-8. The baseline survey was conducted in October-November 2019 (at the beginning of the school year), and the endline survey took place in March-April 2021 (following the end of first semester classes). In 2020, after 3 months of program implementation, program activities were halted from March to October (over 6 months) due to the COVID-19 pandemic, thus the endline survey was postponed to the following school year after implementation was reinitiated.

The overall study objective was to determine the feasibility of delivering adolescent nutrition interventions primarily through school-based platforms and their impact on the diet of adolescent girls.

Research questions include:

1. What is the program impact on the diet of adolescent girls: (1) dietary diversity, (2) meal frequency, and (3) less consumption of unhealthy foods/junk foods?
2. What is the exposure to adolescent nutrition interventions delivered through school-based platforms?
3. What factors influenced the integration of adolescent nutrition interventions into school-based platforms and their outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in primary school grades 4-8
* Parental consent and informed assent received
* Principals, teachers, service providers and primary schools in the areas

Exclusion Criteria:

* Age <10 years or >14 years

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 1712 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Dietary diversity among adolescent girls | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Mean number of food groups consumed by adolescent girls on the day preceding the interview.
Minimum dietary diversity among adolescent girls | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of adolescent girls who consumed 5 or more food groups on the day preceding the interview.

SECONDARY OUTCOMES:
Meal frequency | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Number of meal/snack times in the previous 24 hours
Consumption of unhealthy foods | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Consumption of sweets, baked sweets, sweetened beverages, and fried and salty foods in the previous 24 hours
Exposure to nutrition interventions at school and in the community | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of adolescent girls exposed to nutrition interventions at school and in the community
Nutrition and handwashing knowledge and practices among adolescent girls and their parents | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of adolescent girls and parents with correct knowledge of nutrition and appropriate handwashing practices based on survey responses
Nutrition and handwashing knowledge among school science teachers, principals, and HEWs | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of school science teachers, principals, and HEWs with correct knowledge of nutrition and appropriate handwashing practices based on survey responses
Delivery of adolescent nutrition interventions by school science teachers, principals, and HEWs | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of school science teachers, principals, and HEWs providing adolescent nutrition interventions at school and in the community based on survey responses
Availability of supporting resources | Approximately 17 months after baseline in a cross-sectional endline survey in March-April 2021
  Proportion of primary schools with training and supportive supervision for teachers/staff, educational materials, and healthy food environments based on enumerator observation and survey responses

CONTACTS AND LOCATIONS:
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with donor open access policy requirements, fully anonymized datasets will be made publicly available one year after the end of the project. Metadata and other documentation of data collection procedures (such as the codebook, data collection instruments and interviewer guides/protocols) will also be made publicly available.
Supporting Information: Study Protocol
Time Frame: Fully anonymized datasets will be made publicly available one year after the end of the project.

REFERENCES:
- [Background] Das JK, Salam RA, Thornburg KL, Prentice AM, Campisi S, Lassi ZS, Koletzko B, Bhutta ZA. Nutrition in adolescents: physiology, metabolism, and nutritional needs. Ann N Y Acad Sci. 2017 Apr;1393(1):21-33. doi: 10.1111/nyas.13330. PMID 28436102
- [Background] Spear BA. Adolescent growth and development. J Am Diet Assoc. 2002 Mar;102(3 Suppl):S23-9. doi: 10.1016/s0002-8223(02)90418-9. No abstract available. PMID 11902385
- [Derived] Kim SS, Sununtnasuk C, Berhane HY, Walissa TT, Oumer AA, Asrat YT, Sanghvi T, Frongillo EA, Menon P. Feasibility and impact of school-based nutrition education interventions on the diets of adolescent girls in Ethiopia: a non-masked, cluster-randomised, controlled trial. Lancet Child Adolesc Health. 2023 Oct;7(10):686-696. doi: 10.1016/S2352-4642(23)00168-2. Epub 2023 Sep 1. PMID 37666262

DOCUMENTS (3):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04121559/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04121559/SAP_001.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04121559/ICF_002.pdf